CLINICAL TRIAL: NCT00583661
Title: A Prospective, Multi-center, Single Arm Study to Access the Safety and Probable Benefit of the Berlin Heart EXCOR® Pediatric Ventricular Assist Device [EXCOR Pediatric]
Brief Title: Assess Safety and Probable Benefit of the EXCOR® Pediatric Ventricular Assist Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berlin Heart, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXCOR® Pediatric
Expanded Access: NCT01242891 (Approved for marketing)
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Heart Failure; Cardiomyopathies
Keywords: Ventricular Assist Device; Pediatric Ventricular Assist Device
MeSH Terms: conditions — Heart Failure; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EXCOR Pediatric (Experimental): Implantation of the EXCOR Pediatric Ventricular Assist Device
  Interventions: Device: EXCOR Pediatric

INTERVENTIONS:
Device: EXCOR Pediatric — Extracorporeal Ventricular Assist Device
  Other Names: Berlin Heart; EXCOR®; EXCOR® Pediatric Ventricular Assist Device; EXCOR® Pediatric VAD

SUMMARY:
The purpose of the study is to determine whether use of the Berlin Heart EXCOR® Pediatric Ventricular Assist Device for bridge-to-transplant is associated with a reasonable assurance of safety and probable benefit such that the EXCOR® Pediatric merits approval by the Food and Drug Administration under a Humanitarian Device Exception (HDE).

DETAILED DESCRIPTION:
Berlin Heart Inc. is sponsoring a prospective, multi-center, single arm study to access the safety and probable benefit of the Berlin Heart EXCOR® Pediatric Ventricular Assist Device [EXCOR® Pediatric]. The study will compare the EXCOR® Pediatric with a historical control population supported with extra-corporeal membrane oxygenation (ECMO) as a bridge to cardiac transplantation in children.

ELIGIBILITY:
Inclusion Criteria:

- Severe New York Heart Association (NYHA) Functional Class IV (or Ross Functional Class IV for patients <= 6 years) heart failure refractory to optimal medical therapy, and has met at least one of the following criteria:

* Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) profile status 1 or 1a, i.e. critical cardiogenic shock (low BP unresponsive to support), compromised end organ perfusion, < 24 hour survival without mechanical support; may be due to Ventricular Tachycardia (VT)/Ventricular Fibrillation (VF) (1A) OR
* INTERMACS profile status or 2A (i.e progressive decline): not in imminent danger, but worsening despite optimal inotropic therapy; may be due to VT/VF (2A) AND at least one of the following criteria: Decline in renal functions, Decline in nutritional status, Decline in mobility/ambulation

OR

* Support with extra-corporeal membrane oxygenation (ECMO) or other mechanical circulatory support device OR
* Unable to separate from cardiopulmonary bypass

  * Listed (UNOS status 1A or equivalent) for cardiac transplantation
  * Two-ventricle circulation, including cardiomypathy, repaired structural heart disease or acquired heart disease
  * Age 0 to 16 years
  * Weight >= 3 kg and <= 60 kg
  * Legal guardian (and patient if age-appropriate) understands the nature of the procedure, is willing to comply with associated follow-up evaluations, and provide written informed consent and assent prior to the procedure

Exclusion Criteria:

* Support on ECMO for >= 10 days
* Cardiopulmonary resuscitation (CPR) duration >= 30 minutes within 48 hours of implantation
* Body weight < 3.0 kg or Body Surface Area > 1.5 m2
* Presence of mechanical aortic valve
* Unfavorable or technically-challenging cardiac anatomy including single ventricle lesions, complex heterotaxy, and restrictive cardiomyopathy
* Evidence of intrinsic hepatic disease
* Evidence of intrinsic renal disease
* Evidence of intrinsic pulmonary disease
* Hemodialysis or peritoneal dialysis (not including dialysis or continuous veno-venous hemofiltration (CVVH) for fluid removal)
* Moderate or severe aortic and/or pulmonic valve insufficiency
* Apical Ventricular Septal Defects (VSD) or other compromise that is technically challenging to repair at implant
* Documented heparin induced thrombocytopenia (HIT)
* Documented coagulopathy
* Hematologic disorder
* Active Infection within 48 hours of implant (positive blood culture or White Blood Cell Count >15,000 and fever > 38 degrees C)
* Documented Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)
* Evidence of recent life-limiting malignant disease
* Stroke within 30 days prior to enrollment
* Psychiatric or behavioral disease
* Currently participating in another Investigational Device Exemption (IDE) or Investigational New Drug Application (IND) trial
* Patient is pregnant or nursing

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2007-05; Primary Completion 2010-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles D Fraser, MD, FACS, Principal Investigator — Texas Children's Hospital / Baylor College of Medicine
Locations (17):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Lucille Packard Children's Hospital / Stanford University, Palo Alto, California
  - The Children's Hospital Denver, Denver, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital of Boston, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota - Fairview, Minneapolis, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - The Mt. Sinai Hospital, New York, New York
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Jordan LC, Ichord RN, Reinhartz O, Humpl T, Pruthi S, Tjossem C, Rosenthal DN. Neurological complications and outcomes in the Berlin Heart EXCOR(R) pediatric investigational device exemption trial. J Am Heart Assoc. 2015 Jan 22;4(1):e001429. doi: 10.1161/JAHA.114.001429. PMID 25613996
- [Derived] Fraser CD Jr, Jaquiss RD, Rosenthal DN, Humpl T, Canter CE, Blackstone EH, Naftel DC, Ichord RN, Bomgaars L, Tweddell JS, Massicotte MP, Turrentine MW, Cohen GA, Devaney EJ, Pearce FB, Carberry KE, Kroslowitz R, Almond CS; Berlin Heart Study Investigators. Prospective trial of a pediatric ventricular assist device. N Engl J Med. 2012 Aug 9;367(6):532-41. doi: 10.1056/NEJMoa1014164. PMID 22873533
- [Derived] Almond CS, Buchholz H, Massicotte P, Ichord R, Rosenthal DN, Uzark K, Jaquiss RD, Kroslowitz R, Kepler MB, Lobbestael A, Bellinger D, Blume ED, Fraser CD Jr, Bartlett RH, Thiagarajan R, Jenkins K. Berlin Heart EXCOR Pediatric ventricular assist device Investigational Device Exemption study: study design and rationale. Am Heart J. 2011 Sep;162(3):425-35.e6. doi: 10.1016/j.ahj.2011.05.026. Epub 2011 Jul 30. PMID 21884857
- See also: Berlin Heart Inc. Website — http://www.berlinheart.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject were recruited at pediatric transplant centers by the implanting physicians.
Period: Overall Study
Arm/Group | EXCOR Pediatric
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EXCOR Pediatric
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Median (Full Range); unit: Months] | 64.3 [2.6 to 191.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 47
  Canada | 1

OUTCOME MEASURES:

1. Primary Outcome: The Safety of EXCOR® Pediatric Was Evaluated by Summarizing the Serious Adverse Event Rate Experienced While the Subject Was Supported on the Device.
Description: The serious adverse event rate was calculated by totaling the number of serious adverse events all subjects experienced during device support (from implant to explant, an average of 58 days) divided by the total support time (in days) for all subjects. The serious adverse event rates were calculated separately for each primary study cohort.
Time Frame: Participants were followed while on device support, an average of 58 days
Population: All 48 participants were included in the analysis. Adverse Events for each participant was counted and the total number of events was divided by the total time the Cohort's subjects were supported on device. A 95% Poisson confidence interval was calculated around the point estimates.
Measure: Number (95% Confidence Interval); unit: Events per patient-day
Groups:
- Cohort 1: Subjects with Body Surface Area < 0.7m^2
- Cohort 2: Subjects with Body Surface Area 0.7-1.5m^2
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 24 | 24
Events per patient-day | 0.068 [0.055 to 0.083] | 0.066 [0.053 to 0.081]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2; Ho: EXCOR® SAE Rate >=0.25 Ha: EXCOR® SAE Rate < 0.25 Where serious adverse event (SAE) rate is calculated as the total number of serious adverse events divided by the sum of days all patients are on the EXCOR® Pediatric device, and 0.25 serious adverse events per patient-day is the success criterion. Study success in terms of safety will be demonstrated by the upper bound of a two-sided 95% Poisson exact confidence interval being less than 0.25; Test type: Non-Inferiority or Equivalence — Sample size determination: A sample of 24 subjects followed for approximately 100 days provides greater than 80% power to conclude that, with a 1-sided alpha=0.025 test, the SAE rate of the EXCOR (assumed to be 0.21 per patient-day) is less than 0.25 per patient-day. This sample size was estimated using 10,000 simulations of this study. A total enrollment of 48 subjects (24 per cohort) were enrolled and implanted with the EXCOR® Pediatric; p < 0.05, Poisson confidence interval — A Poisson exact confidence interval was calculated and the critical-value method was used for the significance testing. Success was defined as the upper bound of the 95% Poisson exact confidence interval being less than 0.25; Poisson confidence interval = 0.25, 95% CI 2-sided [0 to 0.25]

2. Primary Outcome: Efficacy of the EXCOR® Pediatric Was Estimated by Showing Survival of All Participants Who Were Supported by the Device.
Description: Efficacy of the EXCOR® Pediatric was estimated by showing survival of all participants who were supported by the device.
Time Frame: Participants were followed while on device support, an average of 58 days
Population: All subjects implanted with the device were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 24 | 24
participants | 21 | 22

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during the time the subject was being supported on the device, an average of 58 days.
Description: Subjects were hospitalized while on device and serious adverse events were assessed on an on-going basis. All reported events were adjudicated by an independent Clinical Events Committee.
Arm/Group | EXCOR Pediatric
Serious Adverse Events (participants affected / at risk) | 41/48
Other Adverse Events (participants affected / at risk) | 3/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EXCOR Pediatric (N=48)
Bleeding (Surgical and medical procedures) | 22 (22)
Cardiac Arrhythmia (Cardiac disorders) | 5 (5)
Pericardial Fluid Collection (Surgical and medical procedures) | 6 (6)
Hemolysis (Blood and lymphatic system disorders) | 2 (2)
Hepatic Dysfunction (Hepatobiliary disorders) | 2 (2)
Hypertension (Cardiac disorders) | 20 (20)
Infection (Infections and infestations) | 27 (27)
Neurological Dysfunction (Nervous system disorders) | 14 (14)
Psychiatric Episode (Psychiatric disorders) | 1 (1)
Renal Dysfunction (Renal and urinary disorders) | 5 (5)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Right Heart Failure (Cardiac disorders) | 5 (5)
Arterial Non-CNS Thromboembolism (Vascular disorders) | 1 (1)
Venous Thromboembolism Event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EXCOR Pediatric (N=48)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI has agreed to discuss or publish trial results only after review by the Publication Committee and the sponsor.